CLINICAL TRIAL: NCT00435357
Title: Comparison Between Fixed- Versus Mobile-bearing TKA : a Randomized Prospective Study
Brief Title: Comparison Between Fixed- Versus Mobile-bearing TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Prof. Philippe NEYRET, Hospices Civils de Lyon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005.407
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Knee Arthritis
Keywords: Mobile-bearing; arthroplasty; fixed-bearing; knee; patella; posterior stabilized TKA
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- mobile-bearing TKA (Experimental)
  Interventions: Device: mobile-bearing TKA
- fixed- bearing TKA (Active Comparator)
  Interventions: Device: fixed- bearing TKA

INTERVENTIONS:
Device: mobile-bearing TKA
  Arms: mobile-bearing TKA
Device: fixed- bearing TKA
  Arms: fixed- bearing TKA

SUMMARY:
The purpose of the study is to analyse the clinical and radiological results of a postero-stabilized TKA by using a mobile bearing versus fixed. Only patients with medial femorotibial arthritis will be included. The consequences on the patellofemoral joint will be thoroughly analysed on skyline view.

ELIGIBILITY:
Inclusion Criteria:

* Medial medial femorotibial arthritis requiring an arthroplasty
* Age between 50y and 90y

Exclusion Criteria:

* Lateral femorotibial arthritis
* Inflammatory disease
* Stiff knee with flexion under 90°
* Revision TKA
* Previous surgery (except meniscectomy)

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
International Knee Society Score | 2, 6 and 12 monthes after surgery

SECONDARY OUTCOMES:
Patellofemoral tilt on skyline view, measurement of two angles : | 2 and 12 monthes after surgery
patellar tilt | 2 and 12 monthes after surgery
patellar displacement from the center of the trochlear groove | 2 and 12 monthes after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Neyret, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Sebastien Lustig, Lyon, France